CLINICAL TRIAL: NCT05729620
Title: Evaluation of STARgraft-3 for Hemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Healionics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP 00530
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: End Stage Renal Disease
Keywords: Hemodialysis; Vascular Access; Arterio-Venous Grafts (AVG)
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- STARgraft-3 (Experimental): Participants will be implanted with 6mm diameter STARgraft-3 grafts as an upper arm Brachial Artery to Axillary Vein shunt for hemodialysis access.
  Interventions: Device: Implant of STARgraft-3 shunt in the upper arm and subsequent use for hemodialysis access

INTERVENTIONS:
Device: Implant of STARgraft-3 shunt in the upper arm and subsequent use for hemodialysis access — After healing from the surgical procedure, the graft will be routinely cannulated for hemodialysis sessions. Periodic evaluations of blood flow by ultrasound imaging will be made over the study period. Established standards of care will be followed as needed to maintain dialysis function.

SUMMARY:
This study is a single site, prospective, single arm evaluation of the safety and effectiveness of the Healionics STARgraft-3 hemodialysis access graft. STARgraft devices have been demonstrated in preclinical and other studies to have improved resistance to the common failure modes of venous anastomosis stenosis and infection.

This study is an extension from prior studies with STARgraft AV (NCT03916731) and STARgraft-2 (NCT04783779) investigational devices. A previous study also included control implants of commercially available standard ePTFE grafts approved for the same use.

The study is enrolling patients with End Stage Renal Disease (ESRD) requiring hemodialysis via a prosthetic vascular graft. The study proposes to evaluate the performance of the investigational STARgraft-3 compared to the ePTFE controls in the prior study and to published results, over a period of 6 months, with extended results to 1 year.

Estimated enrollment is 15 subjects in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, > 18 years or age.
2. Patient has given informed consent to participate in the trial.
3. Stated willingness to comply with all study procedures and availability for the duration of the study.
4. Able to effectively communicate with study personnel.
5. Candidate for a new arterio-venous graft placed in the upper arm.
6. Life expectancy judged to be at least 2 years.
7. Axillary vein of greater than or equal to 7 mm in diameter.
8. Brachial artery of greater than or equal to 4 mm in diameter.
9. Acceptable cardiac risk level (Cardiac Output ≥ 3.5 L/min, Pulmonary Artery Pressure ≤ 50 mmHg, Ejection Fraction ≥ 40%)
10. Systolic blood pressure equal to or greater than 120 mmHg.
11. Absence of central venous stenosis downstream from implant site confirmed with ultrasound and/or venogram.

Exclusion Criteria:

1. Unable or unlikely to comply with trial protocol and/or follow-up.
2. Pregnancy.
3. Clinically morbid obesity.
4. Anatomical limitations.
5. Immunodeficiency syndrome.
6. History of bacterial infection within 8 weeks prior to graft implantation.
7. History of hypercoagulation or bleeding disorders.
8. Elevated platelet count > 1 million per microliter of blood.
9. History of heparin-induced thrombocytopenia syndrome (HIT).
10. Medically confirmed stenosis of the veins downstream of the implant site.
11. Inadequate arterial flow or pressure proximal to the implant site.
12. Currently participating in another investigation drug or device study which may clinically interfere with any endpoints of this trial.
13. Fever greater than 38°C.
14. Prior allergic reaction to silicone.
15. Confirmed or suspected COVID-19 infection within 8 weeks prior to graft implant, or ongoing COVID-19 symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Primary Unassisted Patency | 6 months post implantation
  Percentage of subjects without an occurrence of either an access thrombosis or an access procedure performed to maintain patency.

SECONDARY OUTCOMES:
Primary Unassisted Patency | 1, 2, 4, 9 and 12 months post implantation
  Percentage of subjects without an occurrence of either an access thrombosis or an access procedure performed to maintain patency.
Assisted Primary Patency | 1, 2, 4, 6, 9, and 12 months post implantation
  Percentage of subjects retaining patency after one or more interventions so long as patency was not lost at any point.
Secondary Patency (Cumulative Patency) | 1, 2, 4, 6, 9, and 12 months post implantation
  Percentage of subjects without loss of access at the original implant site.
Frequency of Interventions | 1, 2, 4, 6, 9 and 12 months post implantation
  Frequency of interventions related to graft placement and use for dialysis access.
Blood Flow Rates in Grafts | 2 weeks and 1, 2, 4, 6, 9, and 12 months post implantation
  Ultrasound measurements of flow rates (ml/minute) to detect patency trends with time after implantation.
Safety Outcomes | 1, 2, 4, 6, 9, and 12 months post implantation
  Frequency and severity of Adverse Events resulting from graft implantation and use for hemodialysis access.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Ebner, MD, Principal Investigator — Italian Hospital Asuncion Paraguay
Locations (1):
- Italian Hospital, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: No